CLINICAL TRIAL: NCT05961917
Title: Evaluation of the Effect of Different PEEP Levels on Regional Cerebral Oxygen Saturation in Patients Undergoing Elective Craniotomy for Excision of Brain Tumors ; Randomized Controlled Clinical Trial
Brief Title: Effect of Different Positive End Expiratory Pressures on Regional Cerebral Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halide Hande Şahinkaya, MD, Anesthesiology Specialist, Clinical Director, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NIRS
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Regional Cerebral Oxygen Saturation
Keywords: regional cerebral oxygen saturation; PEEP; craniotomy; near-infrared spectroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group low PEEP (Active Comparator): Positive end-expiratory pressure will be set at 5 cmH2O during controlled mechanical ventilation.
  Interventions: Other: 5 cmH2O Positive end-expiratory pressure (PEEP)
- Group high PEEP (Active Comparator): Positive end-expiratory pressure will be set at 10 cmH2O during controlled mechanical ventilation.
  Interventions: Other: 10 cmH2O Positive end-expiratory pressure (PEEP)

INTERVENTIONS:
Other: 5 cmH2O Positive end-expiratory pressure (PEEP) — PEEP will be set at 5 cmH2O
  Arms: Group low PEEP
Other: 10 cmH2O Positive end-expiratory pressure (PEEP) — PEEP will be set at 10 cmH2O
  Arms: Group high PEEP

SUMMARY:
The goal of this prospective single-blind randomized clinical trial is to compare the effect of two different positive end expiratory pressure (PEEP) levels on regional cerebral oxygen saturation in patients scheduled for craniotomy due to supratentorial masses.

The main question it aims to answer is that how high PEEP level effects the regional cerebral oxygen saturation in patients with high intracranial pressure due to mass effect. Patients will be divided into two groups as Group low PEEP (5 cmH2O) and Group high PEEP (10 cmH2O). Researchers will compare the changes of regional cerebral oxygen saturations between two groups by near infra-red spectroscopy.

DETAILED DESCRIPTION:
In this prospective single-blind study, American Society of Anesthesiologists physical status classification system (ASA) I and II patients aged older than 18 years undergoing craniotomy will be enrolled for the study. Patients will be divided into two groups with computer-based randomization technique. Written and verbal approval will be taken from all patients. Premedication will not be used. Patients will be monitorized by standard non-invasive monitorization (electrocardiography, non-invasive blood pressure measurement, peripheral oxygen saturation) in the operating room. Cerebral/somatic oximeter, near infra-red spectroscopy (NIRS) sensor will be placed on the frontotemporal area and regional cerebral oxygen saturation will be monitorized continuously. Remifentanil infusion with a dose of 0.25 mcg/kg/min will be started two minutes before the induction. After preoxygenation with 6 L/min oxygen for 5 minutes, general anesthesia induction for patients in both groups will be held with intravenous 2 mg/kg propofol. Rocuronium bromide (0.6 mg/kg) will be used for muscle relaxation. Endotracheal intubation will be performed. Controlled mechanical ventilation will be used during the surgery. Invasive arterial blood pressure monitorization will be done and a central venous catheter will be placed in both groups.

In group low PEEP, the patients' settings of mechanical ventilation will be as tidal volume 6-8 mL/kg, inspired oxygen fraction (FiO2) 0.4, PEEP 5 cmH2O. Frequency will be set according to the end tidal carbon dioxide pressure (ETCO2) where it will be 30-32 mmHg.

In group high PEEP, the patients' settings of mechanical ventilation will be as tidal volume 6-8 mL/kg, inspired oxygen fraction (FiO2) 0.4, PEEP 10 cmH2O. Frequency will be set according to the end tidal carbon dioxide pressure (ETCO2) where it will be 30-32 mmHg.

Remifentanil with a dose of 0.05-2 mcg kg/min and propofol with a dose of 50-200 mcg/kg/min will be infused for general anesthesia maintenance in both groups. Dose of remifentanil infusion will be changed according to the blood pressure. If the mean arterial blood pressure and/or heart rate will decrease to 20% of the baseline mean arterial blood pressure and heart rate, the infusion dose will be lowered. If this decrease in heart rate will be over 25%, intravenous 0.5 mg atropin will be administered. If the mean arterial blood pressure will be under 55 mmHg, intravenous 5 mg ephedrine will be administered. If the mean arterial blood pressure will continue to decrease, PEEP will be lowered. If the peripheral oxygen saturation will be under 92%, the inspired oxygen fraction or PEEP will be increased. In these conditions, the patient will be out of study.

1 gr paracetamol will be given intravenously for pain relief. Sugammadex will be used with a dose of 4 mg/kg for extubation.

Regional cerebral oxygen saturation measures will be recorded nine (9) times during the study; pre-induction (period 1), post-induction (period 2), skull pinning (period 3), before dura opening (period 4), after dura opening (period 5), surgical resection of the mass (period 6), dura closure (period 7), end of the surgery (period 8) and end of anesthesia (period 9).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* American Society of Anesthesiologists physical status classification system (ASA) I and II
* Patients scheduled for elective craniotomy
* Patients with supratentorial mass

Exclusion Criteria:

* Hemoglobin concentration lower than 9 mg/dL
* Uncontrolled hypertension
* Congestive heart failure
* Severe chronic obstructive lung disease
* Cerebrovascular disease
* Pulmonary edema
* History of carotis surgery or stenosis of carotid artery
* Unstable hemodynamics
* Pregnancy
* Skin reaction to the NIRS sensor
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
regional cerebral oxygen saturation (SrO2) period 1 | Pre-induction
  The measurement of regional cerebral oxygen saturation before anesthesia induction
regional cerebral oxygen saturation (SrO2) period 2 | Up to 5 minutes after anethesia induction
  The measurement of regional cerebral oxygen saturation after anesthesia induction
regional cerebral oxygen saturation (SrO2) period 3 | From skull-pinning to final head position
  The measurement of regional cerebral oxygen saturation during skull pinning
regional cerebral oxygen saturation (SrO2) period 4 | Just before dura opening
  The measurement of regional cerebral oxygen saturation before dura opening
regional cerebral oxygen saturation (SrO2) period 5 | Up to 5 minutes of dura opening
  The measurement of regional cerebral oxygen saturation after dura opening
regional cerebral oxygen saturation (SrO2) period 6 | During surgical resection
  The measurement of regional cerebral oxygen saturation during surgical resection of the mass
regional cerebral oxygen saturation (SrO2) period 7 | Up to 5 minutes of dura closure
  The measurement of regional cerebral oxygen saturation after dura closure
regional cerebral oxygen saturation (SrO2) period 8 | Within 5 minutes after the surgery
  The measurement of regional cerebral oxygen saturation at the end of surgery
regional cerebral oxygen saturation (SrO2) period 9 | Within 5 minutes after end of anesthesia
  The measurement of regional cerebral oxygen saturation at the end of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Halide H Şahinkaya, MD, Study Chair — University of Health Sciences İzmir Bozyaka Education and Research Hospital; Çağlar Ayar, MD, Study Chair — University of Health Sciences İzmir Bozyaka Education and Research Hospital; Alper Tabanlı, MD, Study Chair — University of Health Sciences İzmir Bozyaka Education and Research Hospital; Zeki T Tekgül, MD, Study Chair — University of Health Sciences İzmir Bozyaka Education and Research Hospital
Locations (1):
- University of Health Sciences İzmir Bozyaka Education and Research Hospital, Izmir, Bozyaka, Turkey (Türkiye)

REFERENCES:
- [Background] Kemerci PU, Demir A, Aydinli B, Guclu CY, Karadeniz U, Cicek OF, Tasoglu I, Ozgok A. 10 cm H2O PEEP application in laparoscopic surgery and cerebral oxygenation: a comparative study with INVOS and FORESIGHT. Surg Endosc. 2016 Mar;30(3):971-8. doi: 10.1007/s00464-015-4277-8. Epub 2015 Jun 23. PMID 26099617
- [Background] Chen H, Zhou XF, Zhou DW, Zhou JX, Yu RG. Effect of increased positive end-expiratory pressure on intracranial pressure and cerebral oxygenation: impact of respiratory mechanics and hypovolemia. BMC Neurosci. 2021 Nov 25;22(1):72. doi: 10.1186/s12868-021-00674-9. PMID 34823465
- [Background] Calderon-Arnulphi M, Alaraj A, Slavin KV. Near infrared technology in neuroscience: past, present and future. Neurol Res. 2009 Jul;31(6):605-14. doi: 10.1179/174313209X383286. PMID 19660190